CLINICAL TRIAL: NCT00335257
Title: International Active Surveillance Study of Women Taking Oral Contraceptives (INAS OC)
Brief Title: International Active Surveillance Study of Women Taking Oral Contraceptives (INAS-OC)
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Juergen Dinger, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG 2005-2
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Contraception
Keywords: Drospirenone; Safety; INAS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Users of OCs containing DRSP
- 2: Users of OCs containing other progestins

SUMMARY:
The study compares the short- and long-term risks of a 24-day regimen of a drospirenone-containing oral contraceptive with the risks of established oral contraceptives in a study population that is representative for the actual users of the individual preparations.

DETAILED DESCRIPTION:
Drospirenone is a novel progestogen with antiandrogenic and antimineralocorticoid properties. A large active post-marketing surveillance study has demonstrated that a 21-day regimen of 3mg drospirenone and 30mcg ethinylestradiol can be used safely for oral contraception. This study investigates the risks of short and long-term use of a 24-day regimen of drospirenone/ethinylestradiol in comparison to established OCs in a study population that is representative of the actual users of the individual preparations.

INAS-OC is a prospective, controlled, non-interventional cohort study with two study arms: OCs containing drospirenone and OCs containing any other progestogen. The study was started in the USA in April 2005 and was extended to several European countries in September 2008 based on the launch status of the 24-day regimen. New users of an OC (starters, switchers without a pill intake break and recurrent users with a pill intake break [same or different OC]) are accrued by a network of prescribing physicians. Baseline and follow-up information are collected via a self-administered questionnaire. Data analysis will be based on life-table methods comparing the cohorts. All analyses will make allowance for confounding, using methods that will include multivariate techniques such as Cox regression.

ELIGIBILITY:
Inclusion Criteria:

* First-ever OC users ("starters")
* Women switching OC use without a pill intake break ("switchers")
* Recurrent users with a pill intake break ("recurrent users")
* Women willing to participate in the active surveillance

Exclusion Criteria:

* Women who do not agree to participate
* Long-term users

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women using oral contraceptives
Sampling Method: Non-Probability Sample
Enrollment: 85109 (Actual)
Dates: Start 2005-08; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen C Dinger, MD, PhD, Principal Investigator — Center for Epidemiology and Health Research, Berlin, Germany
Locations (1):
- Center for Epidemiology and Health Research, Berlin, Germany

REFERENCES:
- [Derived] Dinger J, Bardenheuer K, Heinemann K. Cardiovascular and general safety of a 24-day regimen of drospirenone-containing combined oral contraceptives: final results from the International Active Surveillance Study of Women Taking Oral Contraceptives. Contraception. 2014 Apr;89(4):253-63. doi: 10.1016/j.contraception.2014.01.023. Epub 2014 Feb 4. PMID 24576793
- [Derived] Dinger J, Do Minh T, Buttmann N, Bardenheuer K. Effectiveness of oral contraceptive pills in a large U.S. cohort comparing progestogen and regimen. Obstet Gynecol. 2011 Jan;117(1):33-40. doi: 10.1097/AOG.0b013e31820095a2. PMID 21213475

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 91,474 patients were recruited for the INAS-OC study. Of these, 6,365 participants were excluded due to protocol violations.
Groups:
- OC DRSP-24d: OCs containing DRSP (Yaz®, 24 day regimen)
- OC DRSP-21d: OCs containing DRSP (Yasmin®, 21 day regimen)
- OCs Non-DRSP: Users of OCs containing other progestins
Period: Overall Study
Arm/Group | OC DRSP-24d | OC DRSP-21d | OCs Non-DRSP
Started | 15542 | 9377 | 60190
Completed | 15542 (Numbers completed refer to first follow-up. Individual follow-up ranged between 0.5 and 6.0 years.) | 9377 | 60190 (Numbers completed refer to first follow-up. Individual follow-up ranged between 0.5 and 6.0 years.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- OC DRSP-24d: OCs containing DRSP (Yaz®, 24 day regimen )
- Total: Total of all reporting groups
Arm/Group | OC DRSP-24d | OC DRSP-21d | OCs Non-DRSP | Total
Number analyzed (Participants) | 15542 | 9377 | 60190 | 85109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2054 | 1149 | 7582 | 10785
  Between 18 and 65 years | 13488 | 8227 | 52608 | 74323
  >=65 years | 0 | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.21 (7.64) | 26.14 (7.48) | 26.34 (7.73) | 26.29 (7.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15542 | 9377 | 60190 | 85109
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 922 | 1438 | 11207 | 13567
  United States | 10299 | 3978 | 37892 | 52169
  Austria | 738 | 611 | 2945 | 4294
  Croatia | 509 | 68 | 371 | 948
  Italy | 1644 | 1427 | 2657 | 5728
  Poland | 1169 | 1457 | 3664 | 6290
  Sweden | 261 | 398 | 1454 | 2113

OUTCOME MEASURES:

1. Primary Outcome: Venous Thromboembolism (VTE); Hazard Ratio for DRSP-24 Day vs. Non-DRSP OCs
Description: Venous thromboembolism (VTE) hazard ratio for oral contraceptives containing both drospirenone (DRSP) and ethinylestradiol (EE) in a 24-day regimen or any oral contraceptive without DRSP.
Time Frame: Within 60 months
Population: Study participants that were not excluded due to protocol violation
Measure: Number; unit: participants
Groups:
- OC DRSP-24d: 24-day regimen of DRSP/EE
- OC DRSP-21d: 21-day regimen of DRSP/EE
- OCs Non-DRSP: Users of OCs containing other progestins than DRSP
- NOHC: Non-oral hormonal contraception (injections, implants, levonorgestrel-containing IUDs, or contraceptive patches)
- No Use: No (hormonal) contraception at last contact
Arm/Group | OC DRSP-24d | OC DRSP-21d | OCs Non-DRSP | NOHC | No Use
Number analyzed (Participants) | 7264 | 5605 | 39316 | 4070 | 28854
participants | 19 | 16 | 101 | 7 | 19
Statistical Analysis 1: Comparison: OC DRSP-24d vs OCs Non-DRSP; Tested null hypotheses: the VTE hazard ratio for DRSP(24d) vs. Non-DRSP is higher or equal to 2; Test type: Non-Inferiority or Equivalence — Sample size calculations were based on a non-inferiority test of two exponential survival curves.These calculations are based on the following assumptions: 1) one-sided α 0.025; 2) power (1-β) of 0.90; 3) VTE incidence rate of 9/10.000 WY and 4) non-inferiority limit hazard ratio of 2. Furthermore, a study of this size would exclude a threefold risk of ATE; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.5 to 1.3] — Hazard ratio was adjusted for age, BMI, duration of current use, family history of VTE

2. Primary Outcome: Arterial Thromboembolism (ATE), Hazard Ratio for DRSP-24 Day vs. Non-DRSP OCs
Description: Arterial thromboembolism (ATE) in women using oral contraceptives containing both drospirenone (DRSP) and ethinylestradiol (EE) in a 24-day regimen or any oral contraceptive without DRSP. Cox regression analysis was not carried out. In accordance to the analysis plan, hazard ratios were only to be calculated if a minimum of 5 confirmed events were available in each of the comparison groups.
Time Frame: Within 60 months
Population: Study participants that were not excluded due to protocol violation
Measure: Number; unit: participants
Groups:
- No Use: No (hormonal) contraception
Arm/Group | OC DRSP-24d | OC DRSP-21d | OCs Non-DRSP | NOHC | No Use
Number analyzed (Participants) | 7264 | 5605 | 39316 | 4070 | 28854
participants
  Total number of ATE | 4 | 3 | 30 | 2 | 7
  of which acute myocardial infarction | 2 | 0 | 10 | 1 | 3
  of which ichemic stroke | 1 | 3 | 15 | 0 | 2
  of which transient ischemic attack (TIA) | 1 | 0 | 3 | 0 | 2
  of which peripheral ATE | 0 | 0 | 2 | 1 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected over a time period of 5 years.
Description: Complete cohorts, as-treated population. All study participants were asked for adverse events at each follow-up. The total number of serious adverse events do not include 132 SAEs (due to data entry options), for which information on organ system is missing.
Groups:
- DRSP-24d: 24-day regimen of DRSP/EE
- DRSP-21d: 21-day regimen of DRSP/EE
- NOHC: Non-oral hormonal contraception (injections, implants, levonorgestrel-containing IUDs, or patches)
- No Use: No (hormonal) contraception)
Arm/Group | DRSP-24d | DRSP-21d | OCs Non-DRSP | NOHC | No Use
Serious Adverse Events (participants affected / at risk) | 583/7264 | 499/5605 | 2740/39316 | 254/4070 | 1756/28854
Other Adverse Events (participants affected / at risk) | 0/7264 | 0/5605 | 0/39316 | 0/4070 | 0/28854
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DRSP-24d (N=7264) | DRSP-21d (N=5605) | OCs Non-DRSP (N=39316) | NOHC (N=4070) | No Use (N=28854)
Infectious diseases (Infections and infestations) | 37 | 32 | 137 | 14 | 68
Neoplasms, malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 | 14 | 119 | 7 | 57
Neoplasms, benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5 | 36 | 1 | 14
Diseases of the blood and blood-forming organs (Blood and lymphatic system disorders) | 4 | 5 | 12 | 3 | 15
Endocrine diseases (Endocrine disorders) | 12 | 8 | 47 | 5 | 26
Psychiatric and neurological disorders (Psychiatric disorders) | 53 | 32 | 226 | 23 | 109
Eye (Eye disorders) | 1 | 2 | 14 | 0 | 7
Ear (Ear and labyrinth disorders) | 3 | 7 | 9 | 1 | 6
Cardiovascular system (Cardiac disorders) | 41 | 51 | 278 | 29 | 98
Respiratory system (Respiratory, thoracic and mediastinal disorders) | 39 | 30 | 183 | 18 | 77
Digestive system (Gastrointestinal disorders) | 145 | 116 | 553 | 56 | 259
Skin (Skin and subcutaneous tissue disorders) | 4 | 10 | 40 | 2 | 12
Musculoskeletal system and connective tissue (Musculoskeletal and connective tissue disorders) | 12 | 15 | 81 | 9 | 48
Genitourinary system (Reproductive system and breast disorders) | 93 | 74 | 471 | 44 | 253
Pregnancy, delivery and puerperium (Pregnancy, puerperium and perinatal conditions) | 22 | 32 | 151 | 9 | 571 — SAEs, which occurred within 3 months after stop of hormonal contraceptive use, were attributed to the last OC/NOHC used by the women. Therefore, pregnancy related SAEs in OC/NOHC cohorts do not reflect unwanted pregnancies during OC/NOHC use.
Injury, poisoning, accidents, etc (Injury, poisoning and procedural complications) | 85 | 66 | 383 | 33 | 136

LIMITATIONS AND CAVEATS:
In non-experimental studies the possibility of bias and residual confounding can never be entirely eliminated. The findings may exclude large, but not small relative risks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes